CLINICAL TRIAL: NCT04881929
Title: Study of KN026 in Combination With Docetaxel as Neoadjuvant Therapy in Patients With Early-stage or Locally Advanced HER2-positive Breast Cancer
Brief Title: Study of KN026 in Combination With Docetaxel as Neoadjuvant Therapy in HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN026-208
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN026 + Docetaxel (Experimental): KN026 30 mg/kg IV + Docetaxel 75/m2 every 3 weeks for four cycles
  Interventions: Drug: KN026

INTERVENTIONS:
Drug: KN026 — KN026 in Combination With Docetaxel
  Other Names: Docetaxel

SUMMARY:
This is an open-lable, multicenter, and single arm phase II trial to evaluate treatment with KN026 plus docetaxel as neoadjuvant therapy in patients with early-stage (T1c or 2, N1, M0; T2 or 3, N0, M0) or locally advanced (T1c or 2 or 3, N2, M0; T3N1M0; T1c or 2 or 3, N3a or 3b, M0) HER2-positive breast cancer. The subjects will receive KN026 30 mg/kg IV + Docetaxel 75/m2 every 3 weeks for four cycles prior to surgery.

DETAILED DESCRIPTION:
KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, leading to a dual HER2 signal blockade.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >= 18 years;
* Histologically or cytologically confirmed HER2-positive breast cancer defined as 3+ determined by validated IHC or positive by in situ hybridization (ISH);
* Early-stage (T1c or 2, N1, M0; T2 or 3, N0, M0) or locally advanced (T1c or 2 or 3, N2, M0; T3N1M0; T1c or 2 or 3, N3a or 3b, M0) breast cancer;
* Adequate organ function assessed within 7 days prior to first trial treatment;
* ECOG score 0 or 1;
* Left ventricular ejection fraction (LVEF) ≥ 55% at baseline;

Exclusion Criteria:

* Stage IV (metastatic) breast cancer;
* Inflammatory breast cancer;
* Previous anti-cancer therapy or radiotherapy for any malignancy;
* Major surgery for any reason within 28 days;
* History of uncontrolled intercurrent illness;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
tp CR as assessed by local pathologist | up to 12 weeks
  total pathological complete response as assessed by local pathologist

SECONDARY OUTCOMES:
bp CR as assessed by local pathologist | up to 12 weeks
  breast pathological complete response assessed by local pathologist
ORR as assessed by the investigator according to RECIST 1.1 | up to 12 weeks
  Objective response rate as assessed by the investigator according to RECIST 1.1
safety as assessed by the investigator according to RECIST 1.1 | up to 12 weeks
  Incidence, type, and severity of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No